CLINICAL TRIAL: NCT03478215
Title: A Double-blind, Randomized, Controlled Dose Escalation Trial of Autologuous Mesenchymal Stromal Cells in Living Donor Kidney Transplant Recipients
Brief Title: Mesenchymal Stromal Cells in Living Donor Kidney Transplantation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Ahmed Osama Gaber, MD, Principal Investigator, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Pro00012858; U1111-1169-2289 (Other: Universal Trial Number)
Record Dates: First submitted 2016-03-18; First posted 2018-03-27 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Renal Transplantation; Mesenchymal Stem Cells
Keywords: kidney transplantation; graft rejection
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mesenchymal Stromal Stem Cells Infusion (Experimental): Intervention: Mesenchymal stromal stem cells infusion. This is the active investigational intervention, administered intravenously at surgery and day 4 post-transplant in a dose-escalation fashion beginning as 1x10^6 cells for the first dose group, 2x10^6 cells for the second dose group, or 3x10^6 cells for the last dose group. The infusion set-up will be covered to mask the group assignment.
  Participants will also receive BASILIXIMAB (Simulect, for all subjects at a standard dose, 20mg reconstituted with normal saline or 5% dextrose) on the day of surgery and day 3 or 4 post-transplant administered by a member of the anesthesia team; TACROLIMUS (Prograf for maintenance therapy), MYCOPHENOLATE MOFETIL (Cellcept for maintenance therapy), and CORTICOSTEROIDS as routine care.
  Interventions: Biological: Mesenchymal Stromal Stem Cells (MSCs) Infusion
- Placebo Infusion (Placebo Comparator): Placebo: A normal saline infusion. This is the placebo intervention to occur at surgery and day 4 post-transplant. The infusion set-up will be covered to mask the group assignment. Participants will also receive BASILIXIMAB (Simulect, for all subjects at a standard dose, 20mg reconstituted with normal saline or 5% dextrose) on the day of surgery and day 3 or 4 post-transplant administered by a member of the anesthesia team; TACROLIMUS (Prograf for maintenance therapy), MYCOPHENOLATE MOFETIL (Cellcept for maintenance therapy), and CORTICOSTEROIDS as routine care.
  Interventions: Other: Normal Saline (Placebo) Infusion

INTERVENTIONS:
Biological: Mesenchymal Stromal Stem Cells (MSCs) Infusion — Investigational infusion bag containing autologous mesenchymal stromal cells wrapped to cover contents to maintain the blind.
  Mesenchymal Stromal Stem Cells Infusion.
  Other Names: Investigational autologous biological product
  Arms: Mesenchymal Stromal Stem Cells Infusion
Other: Normal Saline (Placebo) Infusion — Matching infusion containing normal saline wrapped to cover contents to maintain the blind.
  Normal Saline (Placebo) Infusion.
  Other Names: Matching placebo infusion bag
  Arms: Placebo Infusion

SUMMARY:
Kidney transplantation is a good treatment option for people with kidney disease. However, there is still much to learn about how to best care for the transplanted kidney and keep it functioning for a long time. Transplant recipients receive induction therapy and immunosuppression (anti-rejection) drugs to prevent their body from rejecting the new kidney. These drugs are used to prevent the immune system from attacking the transplanted kidney. This research study will evaluate the safety and activity of mesenchymal stromal stem cells (MSCs) infusion compared to saline-only infusion in reducing the immune suppression necessary to achieve optimal renal function in renal transplant recipients. All participants will receive routine care: basiliximab, tacrolimus, mycophenolate mofetil, and corticosteroids.

DETAILED DESCRIPTION:
The study is a double-blind, randomized, controlled, dose-escalation and safety study of the investigational product, autologous MSCs, to be assessed for inducing immune suppression in living donor kidney transplant recipients as compared to saline, the placebo infusion. The investigator will obtain exploratory immune response markers to estimate the effect of autologous MSCs on the T- and B-cell response following living donor kidney transplantation. The usual routine care supportive drugs will be given to all: corticosteroids during induction, the calcineurin inhibitor tacrolimus (Prograf®, Astellas Pharma), and mycophenolate mofetil (Cellcept®, Genentech) for maintenance therapy. All subjects will receive basiliximab (Simulect®, Novartis), a standard drug used to induce immune suppression.

Up to 24 patients will be enrolled at the Houston Methodist Hospital. Safety analyses will be conducted after the first 4 subjects have been enrolled and completed the first 30-90 days posttransplant, with subject 2 enrolled 30 days after subject 1 and subject 3 enrolled 30 days after subject 2 (eg, a 30-day window between subject enrollment days). If no safety signal has been detected, the next group of 4 subjects will be enrolled using no less than a 2-week enrollment window from subject 5, 2 weeks from subject 6, and so on. Subjects will be evaluated in the same manner until 8 subjects in the final dosing group have completed 90 days or a decision to stop the study has occurred, whichever comes first. Each subsequent dosing group will begin with a 30-day window of evaluation between subjects enrolled for the first 4 subjects enrolled in the group. If no adverse safety signal has been detected in the first 4 cases in that dosing group, the next 4 subjects enrolled will have a 2-week evaluation window between enrollments. This early evaluation approach will allow for the assessment of the inflammatory period occurring after transplantation. A final safety review will occur at the end of the study and a report will be written.

The study will provide information needed to select a MSC dose level to be used in subsequent clinical trials and to inform the design of subsequent trials.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females from 18 to 65 years of age
2. Planned to receive a primary kidney transplant from a living donor
3. Low immunologic risk defined as

   1. No history of current or historical antidonor human leukocyte antigen (HLA) antibodies (DSA)
   2. Panel of Reactive Antibodies (PRA) <20%, historical
4. Low risk for thrombotic events and normal prothrombin time, international normalized ratio (INR) and partial thromboplastin time
5. Women of child bearing potential have a negative serum pregnancy test prior to transplantation
6. Women of child bearing potential (including perimenopausal women who have had a menstrual period within the previous 1 year) who agree to use 2 forms of effective birth control regimen (at least one of which is a barrier method) throughout the study period and for 6 weeks following the end of the study or the last dose of mycophenolate mofetil, whichever comes first.
7. In the opinion of the investigator, the subject is capable of understanding and complying with the protocol.
8. Subjects must have signed the informed consent document prior to performance of any study related procedure including screening procedure.

Exclusion Criteria:

1. Recipient of multiple organ transplantation or scheduled for multiple organ transplantation
2. Recipient with a donor-specific anti-HLA antibody or positive cross-match requiring deviation from standard immunosuppressive therapy
3. Hepatitis C antibody positive, Hepatitis B antigen positive, or Hepatitis B core antibody positive
4. Currently participating in or has participated in an investigational drug or medical device study within 30 days or five half-lives, whichever is longer, prior to enrollment into this study
5. Concurrent sepsis or active bacterial infection
6. In the opinion of the investigator is anatomically a high-risk renal transplant with higher chance for thrombosis or bleeding
7. Have an active malignancy or history of solid, metastatic or hematologic malignancy with the exception of basal or squamous cell carcinoma of the skin that has been treated
8. Women of child bearing potential who are breastfeeding
9. History of HIV infection
10. Subject is unwilling or unable to comply with the protocol or to cooperate fully with the Investigator or the site personnel.
11. Subject is not deemed medically stable for the study in the opinion of the Investigator or the subject's nephrologist.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants without any infusional toxicity, occurring within 24 hours of infusion. | 24 hours from end of infusion
  Infusional toxicity will be assessed as the occurrence of either 1) two or more participants having deep vein thrombosis (Grade 2 thrombotic event); 2) any participant having evidence of the first-pass phenomenon of cells trapping in the lung as evidenced by (a) shortness of breath at rest, (b) requiring ventilator support, or (c) pulmonary edema with hypoxia requiring support; or 3) Grade 4 hypertension or hypotension; or 4) acute myocardial infarction; or 5) new onset congestive heart failure; or 6) capillary leak syndrome; or 7) acute kidney injury; or 8) biopsy-proven rejection.

SECONDARY OUTCOMES:
Number of participants without any acute rejection, graft loss, or death at 6 months post transplant. | 6 months post transplant
  Rejection will be determined as biopsy-proven allograft rejection (BPAR). Graft loss will be counted when the patient loses kidney function to the point that they require chronic renal replacement therapy (e.g., dialysis for more than 8 weeks or a re-transplant).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed O Gaber, MD, Principal Investigator — Houston Methodist Physicians Organization
Locations (1):
- Houston Methodist Hospital System, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No